CLINICAL TRIAL: NCT07189572
Title: Efficacy of Intranasal Corticosteroid Spray in Preventing Otitis Media With Effusion After Radiotherapy for Nasopharyngeal Carcinoma: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase III Clinical Trial
Brief Title: Intranasal Corticosteroid Spray for Preventing Otitis Media With Effusion After Radiotherapy in Nasopharyngeal Carcinoma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Sun Yat-sen University (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UHCT250873
Record Dates: First submitted 2025-09-16; First posted 2025-09-24 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Otitis Media; Otitis Media With Effusion After Nasopharyngeal Carcinoma; Radiotherapy Side Effects; Radiotherapy Side Effect; Otitis Media With Effusion (OME)
MeSH Terms: conditions — Otitis Media; Radiation Injuries; Otitis Media with Effusion | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Triamcinolone Acetonide Nasal Spray (Experimental): Participants will receive triamcinolone acetonide nasal spray (55 μg/spray) in addition to concurrent cisplatin-based chemoradiation. The intervention is initiated on day 1 of radiotherapy. The dosing regimen is 2 sprays per nostril (total daily dose of 220 μg) administered each morning for 12 weeks, covering the entire radiotherapy course and the acute inflammatory phase. All patients will also perform daily nasal irrigation with normal saline, timed at least 30 minutes apart from the drug administration.
  Interventions: Drug: Triamcinolone Acetonide
- Placebo Nasal Spray (Placebo Comparator): Participants will receive a matching placebo nasal spray, which is identical in appearance and usage to the active drug, in addition to concurrent cisplatin-based chemoradiation. The intervention is initiated on day 1 of radiotherapy. The dosing regimen is 2 sprays per nostril administered each morning for 12 weeks. All patients will also perform daily nasal irrigation with normal saline, timed at least 30 minutes apart from the placebo administration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Triamcinolone Acetonide — Triamcinolone acetonide is a medium-potency synthetic corticosteroid. This intervention is administered via a commercially available, metered-dose nasal spray that delivers 55 μg of the active drug per spray. It exerts potent local anti-inflammatory and immunomodulatory effects in the nasal mucosa and Eustachian tube orifice. In this study, it is investigated for the prevention of radiotherapy-induced otitis media with effusion in patients with nasopharyngeal carcinoma.
  Arms: Triamcinolone Acetonide Nasal Spray
Drug: Placebo — The placebo nasal spray is specifically formulated to be indistinguishable from the active triamcinolone acetonide nasal spray. It is identical in all physical properties including appearance, scent, taste, packaging, and administration procedure. It contains the same inactive excipients (e.g., preservatives, suspending agents) but does not contain any triamcinolone acetonide or other active pharmaceutical ingredient.
  Arms: Placebo Nasal Spray

SUMMARY:
This study focuses on a common side effect experienced by many patients after radiation therapy for nasopharyngeal cancer, which is a type of head and neck cancer. This side effect is called secretory otitis media (fluid buildup in the middle ear). It can cause a feeling of fullness in the ear and hearing loss. While procedures like ear tube placement can help, they can also lead to other problems like ear infections and drainage.

Radiation treatment is thought to cause inflammation that disrupts the normal function of the tube connecting the ear to the throat (Eustachian tube), leading to this fluid buildup. A nasal spray containing a steroid medicine (triamcinolone acetonide) is already known to be safe and effective at reducing inflammation in the ear fluid of both children and adults. We believe that using this spray may also help prevent and improve this condition in nasopharyngeal cancer patients after radiation therapy.

The main goal of this study is to explore whether this nasal spray can effectively prevent or reduce fluid buildup in the ear following radiation therapy. We hope this non-invasive treatment will provide a new option to improve the quality of life for these patients.

DETAILED DESCRIPTION:
Background and Rationale:

Nasopharyngeal carcinoma (NPC) is endemic in Southern China. While radiotherapy has significantly improved survival rates, radiation-induced complications severely impact quality of life. Otitis media with effusion (OME) is a highly prevalent complication, with an acute phase (during radiotherapy up to 3 months post-treatment) incidence of 30%-70%. Notably, 20%-40% of these cases progress to chronic OME, and 10%-30% require invasive procedures like tympanostomy tube insertion due to persistent symptoms and hearing loss (often >30 dB).

The pathophysiology of radiation-related OME is distinct from generic OME. It involves mucosal injury in the Eustachian tube region (especially at radiation doses ≥60 Gy), leading to ciliary dysfunction, local immune dysregulation, and mechanical obstruction. Post-radiation changes also include mucosal structure alteration, local immunosuppression, and impaired mucociliary clearance, creating a persistent inflammatory environment conducive to effusion formation.

Current management, primarily adapted from conventional OME protocols (e.g., tympanostomy), offers short-term symptom relief but is associated with significant long-term complications, including chronic otorrhea (15%-20%) and persistent tympanic membrane perforation (5%-10%). This highlights the critical need for preventive and non-invasive strategies targeting the underlying inflammatory etiology.

Topical intranasal corticosteroids, such as triamcinolone acetonide, offer a mechanistically grounded prophylactic approach. They exert potent local anti-inflammatory and immunomodulatory effects by targeting and inhibiting the NF-κB pathway. This action can potentially mitigate mucosal inflammation, restore ciliary function, and rebalance local immunity in the nasopharynx and Eustachian tube orifice during and after radiotherapy, thereby preventing the initiation of the effusion process. Evidence supports their efficacy and safety in managing OME in other populations, with randomized controlled trials (e.g., by El-Anwar et al.) showing non-inferiority to systemic steroids with a significantly improved adverse effect profile (60%-70% reduction in systemic adverse events), making them suitable for long-term use in this patient population.

Study Objective and Design:

This study is a phase III, multicenter, randomized, double-blind, placebo-controlled trial designed to evaluate the efficacy of prophylactic intranasal triamcinolone acetonide in reducing the incidence and severity of radiation-related OME in patients with NPC.

The intervention will be initiated concurrently with radiotherapy. Participants will be randomly assigned to receive either triamcinolone acetonide nasal spray or an identical placebo spray. The primary outcome is the incidence of clinically significant OME requiring intervention within a specified post-radiation period. Key secondary endpoints include objective measures of hearing function (pure-tone audiometry to assess hearing threshold shifts), tympanometric changes, the need for invasive procedures (tympanocentesis or tube placement), and patient-reported quality of life measures assessed using validated questionnaires.

This study aims to provide high-level evidence for a novel, preventive strategy targeting the inflammatory pathogenesis of radiation-induced OME, ultimately aiming to improve long-term otological outcomes and quality of life for NPC survivors.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed nasopharyngeal carcinoma scheduled for curative intensity-modulated radiation therapy (IMRT), with or without concurrent chemotherapy.
* Age between 18 and 75 years.
* No previous history of head and neck radiotherapy.
* Intact tympanic membranes bilaterally at baseline, with no history of middle ear surgery (including tympanostomy tube placement).
* Willing to comply with all study procedures, including nasal spray use, audiological examinations, and follow-up visits.
* No use of systemic or topical corticosteroids, antihistamines, or decongestants within 14 days prior to randomization.
* All inclusion criteria must be met for participation

Exclusion Criteria:

* Diagnosed with complete conductive hearing loss or ossicular chain fixation.
* Scheduled to undergo tympanostomy tube placement, tympanotomy, or other middle ear surgery prior to randomization.
* Unlikely to complete the 12-month follow-up (e.g., planned relocation, poor compliance).
* Presence of respiratory conditions requiring treatment with nasal corticosteroids.
* Known allergy or hypersensitivity to nasal corticosteroids (especially triamcinolone acetonide or its excipients).
* History of severe mental illness, cognitive impairment, or substance abuse that may affect compliance.
* Pregnant or lactating women, or women of childbearing potential unwilling to use effective contraception.
* Participation in other investigational drug clinical trials within the past 3 months.
* Deemed unsuitable for the trial by the investigator (e.g., severe septal deviation, chronic rhinosinusitis requiring systemic treatment, or poorly controlled diabetes).
* Any subject who meets any of the above exclusion criteria at baseline will be excluded from the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of Otitis Media with Effusion (OME) within 12 months after radiotherapy | From initiation of study intervention (radiotherapy start) until 12 months after completion of radiotherapy.
  The occurrence of OME is determined by a combination of: 1) Presence of relevant symptoms (e.g., ear fullness, hearing loss); AND 2) Confirmatory physical examination findings on otoscopy (e.g., tympanic membrane retraction, air-fluid levels, bubbles); AND 3) Objective evidence from tympanometry (Type B or Type C curve, indicating middle ear effusion or significant negative pressure). A case of OME is only confirmed if all three criteria are met. The incidence is calculated as the proportion of participants in each group who develop confirmed OME at any point during the 12-month follow-up period after the completion of radiotherapy.

SECONDARY OUTCOMES:
Time to onset of Otitis Media with Effusion (OME) | From the start of radiotherapy until the first occurrence of OME, assessed up to 12 months after radiotherapy completion.
  This measures the time from the start of radiotherapy (baseline) to the first diagnosis of OME. Diagnosis requires the concurrent presence of: 1) relevant symptoms (e.g., ear fullness, hearing loss); 2) confirmatory findings on otoscopy; and 3) a Type B or C tympanogram. The time-to-event data will be analyzed using methods such as Kaplan-Meier curves and Cox proportional hazards models to compare the difference between study arms. Additionally, the proportion of participants with early-onset OME (within 1 month post-radiotherapy) and late-onset OME (after 3 months post-radiotherapy) will be compared between groups using chi-square tests.
Change in pure-tone average hearing threshold | Baseline (pre-radiotherapy), and at 3 month, 6 months, and 12 months after completion of radiotherapy.
  Hearing function is assessed by pure-tone audiometry. The pure-tone average (PTA) will be calculated for low frequencies (500 Hz), medium frequencies (1000, 2000 Hz), and high frequencies (4000 Hz). Change from baseline (pre-radiotherapy) in PTA at each post-treatment timepoint will be calculated and compared between groups. The incidence of clinically significant hearing loss, defined as a threshold shift of ≥15 dB HL at the affected frequencies, will also be compared. The severity of hearing loss will be categorized based on PTA as mild (26-40 dB HL), moderate (41-60 dB HL), or severe (>60 dB HL).
Tympanometry results | Baseline (pre-radiotherapy), and at 3 month, 6 months, and 12 months after completion of radiotherapy.
  Middle ear function is assessed by tympanometry. Results will be categorized according to standard Jerger classification: Type A (normal), Type B (flat, suggesting effusion), and Type C (negative pressure, suggesting Eustachian tube dysfunction). The distribution of tympanogram types, actual tympanometric peak pressure values (in daPa), and static acoustic compliance values (in mL) will be compared between groups at each timepoint. The primary focus is on the incidence of abnormal tympanograms (Type B or C). Additionally, the conversion rate from an abnormal tympanogram to a normal Type A tympanogram will be analyzed as a measure of recovery.
Change in disease-specific quality of life scores | Baseline (pre-radiotherapy), and at 3 months, 6 months, and 12 months after completion of radiotherapy.
  Description [*] The impact on quality of life is assessed using two validated patient-reported outcome measures: the EORTC QLQ-H&N35 module (specific to head and neck cancer patients) and the ETDQ-7 questionnaire (specific to Eustachian tube dysfunction). The QLQ-H&N35 assesses symptoms and social function, while the ETDQ-7 focuses on ear-related symptoms. Change scores from baseline for each questionnaire will be calculated. A decrease in the score represents an improvement in symptoms and quality of life. The mean change in scores at each post-radiotherapy timepoint will be compared between the two study arms.